CLINICAL TRIAL: NCT03892642
Title: Phase Ib Study of Avelumab Plus Bacille Calmette-Guerin (BCG) in Patients With Non-muscle Invasive Bladder Cancer (ABC Trial)
Brief Title: Avelumab Plus Bacille Calmette-Guerin (BCG) in Patients With Non-muscle Invasive Bladder Cancer
Acronym: OU-SCC-ABC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-ABC; OU-SCC-ABC (Other Grant/Funding Number: EMD Serono)
Record Dates: First submitted 2019-02-07; First posted 2019-03-27 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Bladder Cancer
Keywords: Intravesical BCG; Bacille Calmette-Guerin; avelumab
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BCG + Avelumab (Experimental): Combination of avelumab and intravesical BCG. One cycle = 12 weeks (84 days). A standard maintenance therapy regimen will be provided with BCG occurring at Month 3, 6, and 12. Avelumab treatment ends at the conclusion of Month 12 maintenance therapy.
  Interventions: Drug: Avelumab; Biological: BCG

INTERVENTIONS:
Drug: Avelumab — Induction phase:
  * once weekly for weeks 1-6,
  * once every 2 weeks at week 8, 10, and 12
  Maintenance phase:
  * Once every week for weeks 1-3
  * Once every 2 weeks starting at week 5, until the next BCG treatment
Biological: BCG — Induction phase (cycle 1):
  • Once weekly for weeks 1-6
  Maintenance phase (Month 3, 6, and 12):
  • Once weekly for 3 weeks
  Other Names: Bacille Calmette-Guérin

SUMMARY:
The purpose of this study is to test the safety of avelumab and Bacille Calmette-Guerin (BCG) and see what effects (good and bad) that this combination treatment has on subjects with recurrent bladder cancer.

DETAILED DESCRIPTION:
There will be exams, tests and procedures to see if the patient is eligible for the study. Some are part of regular cancer care and others are part of the study. Subjects will also need to complete a research questionnaire at certain points in the study.

Subjects will receive treatment of avelumab and intravesical BCG until unacceptable toxicity or tumor progression.

Study participation is up to three years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented Non-muscle Invasive Bladder Cancer (NMIBC)
2. Patient with BCG-treated but unresponsive NMIBC (persistent or recurrent defined as tumor lesion present after prior response).
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 2.
4. Patients who are able to understand and sign the informed consent form.
5. Age ≥ 18 years old
6. Ability to comply with protocol
7. Life expectancy >/=12 weeks
8. Adequate hematologic and end-organ function per protocol
9. For women of childbearing potential: Negative serum or urine pregnancy test at screening.
10. For both male and female subjects: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 30 days after the last dose of study drug.

Exclusion Criteria:

1. Evidence of locally advanced or metastatic bladder cancer (including current disease involving renal pelvis, ureter, or prostatic urethra).
2. Evidence of muscle-invasive bladder cancer
3. Evidence of extravesical bladder cancer
4. Active central nervous system (CNS) metastases.
5. Prior treatment with PD-L1 or PD-1 inhibitor.
6. Prior radiation to bladder
7. Known additional malignancy that required active treatment within the last 2 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin.
8. Patient is considered a poor medical risk that would interfere with cooperation with the requirements of the study.
9. Patient has a condition or laboratory abnormality that might confound the study results, or interfere with the patient's participation for the full duration of the study treatment.
10. Patient has not recovered (i.e, to ≤Grade 1 or to baseline) from previous intravesical BCG or other anti-cancer therapy induced AEs.
11. Treatment with any approved anti-cancer therapy, including chemotherapy (systemic or intravesical), radiation therapy, or hormonal therapy within 3 weeks prior to the first dose of study treatment
12. Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 4 weeks prior to the first dose of study treatment
13. Pregnant or lactating, or intending to become pregnant during the study

    a. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to the first dose of study treatment.
14. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
15. Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells
16. Allergy or hypersensitivity to components of the avelumab formulation
17. History of autoimmune disease defined per protocol
18. Prior allogeneic stem cell or solid organ transplantation
19. Current use of immunosuppressive medication defined per protocol
20. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan

    a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
21. Positive test for HIV
22. Active hepatitis B (positive hepatitis B surface antigen [HBsAg] test at screening);

    a. Patients with past or resolved hepatitis B (HBV) infection (positive anti-hepatitis B core antigen [anti-HBc] antibody test) are eligible. HBV DNA must be obtained in these patients prior to the first dose of study treatment.
23. Active hepatitis C

    a. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction assay is negative for HCV RNA.
24. Active infection requiring systemic therapy
25. Severe infections within 4 weeks prior to the first dose of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
26. Significant cardiovascular disease, such as cerebral vascular accident/stroke (< 6 months prior to enrollment), New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina
27. Administration of a live/attenuated vaccine within 4 weeks prior to the first dose of study treatment, within 5 months following the administration of the last dose of study drug, or anticipation that such a live/attenuated vaccine will be required during the study
28. Other severe acute or chronic medical conditions defined per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2023-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Stratton, MD, Principal Investigator — Stephenson Cancer Center
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the Stephenson Cancer Center began in May 2019, with the first patient consenting, and last patient consent occurred in February 2021. The Stephenson Cancer is no longer recruiting for this study as all the slots have been filled and subjects accrued per protocol.
Groups:
- BCG + Avelumab: Combination of avelumab and intravesical BCG. One cycle = 12 weeks (84 days). A standard maintenance therapy regimen will be provided with BCG occurring at Month 3, 6, and 12. Avelumab treatment ends at the conclusion of Month 12 maintenance therapy.
  Avelumab: Induction phase:
  * once weekly for weeks 1-6,
  * once every 2 weeks at week 8, 10, and 12
  Maintenance phase:
  * Once every week for weeks 1-3
  * Once every 2 weeks starting at week 5, until the next BCG treatment
  BCG: Induction phase (cycle 1):
  • Once weekly for weeks 1-6
  Maintenance phase (Month 3, 6, and 12):
  • Once weekly for 3 weeks
Period: Overall Study
Arm/Group | BCG + Avelumab
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who enrolled in study
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.94 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Receiving Complete Induction Course
Description: Proportion of patients receiving complete induction course, defined as freedom from DLT preventing completion of at least 5 of 6 treatments of BCG + avelumab
Time Frame: 8 weeks
Population: Patients who enrolled in study
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 18
proportion of patients | 0.833 [0.5774 to 0.9559]

2. Secondary Outcome: Proportion of Patients Receiving Complete Induction Course
Description: completion of at least 2 of 3 treatments within each 5 week period
Time Frame: 5 weeks
Population: Patients who remained on study for induction course
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 11
proportion | 0.9091 [0.5712 to 0.9952]

3. Secondary Outcome: Percent of Patients With Complete Response
Description: based on negative cystoscopy and urine cytology. A negative biopsy at 6 months will provide evidence of complete response.
Time Frame: 3 months
Population: Patients who enrolled in study
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 18
percent of patients | 17.6 [3.8 to 43.4]

4. Secondary Outcome: Proportion of Patients With Complete Response
Description: as for outcome 3
Time Frame: 6 months
Population: Patients who enrolled in study
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 18
percent | 41.2 [18.4 to 67.1]

5. Secondary Outcome: Percent of Patients With Recurrence Free Survival
Description: defined as percent of patients who are alive and free of persistent or recurrent NMIBC based on cystoscopy, cytology and/or biopsy.
Time Frame: 6 months
Population: Patients who experienced complete response
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 9
percent of patients | 88.89 [43.29 to 98.36]

6. Secondary Outcome: Proportion of Patients With Recurrence Free Survival
Description: defined as proportion of patients who are alive and free of persistent or recurrent NMIBC based on cystoscopy, cytology and/or biopsy
Time Frame: 12 months
Population: Patients who experienced complete response
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 9
proportion of patients | 0.8889 [.4329 to .9836]

7. Secondary Outcome: Proportion of Patients With Progression-free Survival
Description: defined by time from day of first treatment to first progression to higher grade or stage, including muscle-invasive disease or death from any cause
Time Frame: 6 months
Population: Patients who experienced progression or death or who stayed on study for at least 6 months
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 17
proportion of patients | 0.8824 [.6059 to .9692]

8. Secondary Outcome: Proportion of Patients With Progression-free Survival
Description: as for outcome 7
Time Frame: 12 months
Population: Patients who experienced progression or death or who remained at study at least 12 months
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | BCG + Avelumab
Number analyzed (Participants) | 15
proportion of patients | 0.8145 [.5263 to .9364]

ADVERSE EVENTS:
Time Frame: 2 years, 9 months
Description: AEs graded according to CTCAE v 5.0
Arm/Group | BCG + Avelumab
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 11/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCG + Avelumab (N=18)
Atrial flutter (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Cardiac troponin I increased (Investigations) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCG + Avelumab (N=18)
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Other SpecifyDiverticulitis (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 6
Flu like symptoms (General disorders) | 4
Infusion site extravasation (General disorders) | 1
Penile infection (Infections and infestations) | 1
Shingles (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 7
Bruising (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 5
Activated partial thromboplastin time prolonged (Investigations) | 1
CPK increased (Investigations) | 2
Cardiac troponin I increased (Investigations) | 1
Creatinine increased (Investigations) | 4
Thyroid stimulating hormone increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Psychiatric disorders) | 1
Bladder spasm (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 11
Hematuria (Renal and urinary disorders) | 5
Other SpecifyNOCTURIA (Renal and urinary disorders) | 1
Other SpecifyUrinary Disorder (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 10
Urinary retention (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 5
Other Specify (Reproductive system and breast disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Prostatic pain (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT03892642/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT03892642/SAP_001.pdf